CLINICAL TRIAL: NCT05141435
Title: NHFOV vs nCPAP in Very Preterm Infants With Respiratory Distress Syndrome: A Multi-center, Prospective, Randomized, Controlled Clinical Superior Trial
Brief Title: NHFOV as Primary Support in Very Preterm Infants With RDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiulongpo No.1 People's Hospital (Other)
Collaborators: Jiangxi Maternal and Child Health Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Guiyang Maternity and Child Health Care Hospital (Other); The Second Hospital of Shandong University (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Women and Children's Health Hospital of Yulin (Other); Chongqing Three Gorges Central Hospital (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); The First People's Hospital of Yunnan (Other); Chengdu Women's and Children's Central Hospital (Other); Maternal and Children's Healthcare Hospital of Taian (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Quanzhou Children's Hospital (Other); Chongqing West Hospital (Other); Chongqing Medical Center for Women and Children (Other); Xiamen Maternity & Child Care Hospital (Other); Qujing Maternal and Child Health Hospital (Other); Liuzhou Maternity and Child Healthcare Hospital (Other); International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Xingwang Zhu, Doctor, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHFOV prevent intubation
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: to Test the Hypothesis That NHFOV is More Effective Than nCPAP in the Treatment of Respiratory Distress Syndrome (RDS) in Verypreterm Neonates
Keywords: nasal high frequency oscillation ventilation(NHFOV); nasal continuous positive airway pressure(NCPAP); preterm infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCPAP (Active Comparator)
  Interventions: Procedure: infants receive primary non-invasive respiratory support by mean of nCPAP; Procedure: infants receive primary non-invasive respiratory support by mean of NHFOV
- NHFOV (Active Comparator)
  Interventions: Procedure: infants receive primary non-invasive respiratory support by mean of nCPAP; Procedure: infants receive primary non-invasive respiratory support by mean of NHFOV

INTERVENTIONS:
Procedure: infants receive primary non-invasive respiratory support by mean of nCPAP — neonates assigned to the nCPAP group will be started on a pressure of 6 cmH2O( adjust range:6-10 cmH2O) , with FiO2 (0.21-0.40)adjusted to target SpO2 from 89% to 94%. CPAP will be provided by either variable flow or continuous flow devices, as there is no clear evidence that one type of CPAP generator would be better than any other by pure CPAP system.
Procedure: infants receive primary non-invasive respiratory support by mean of NHFOV — neonates assigned to NHFOV will be started with the following boundaries: a) Paw of 6 cmH2O (the range 6-10 cmH2O); b) frequency of 10 Hz (the range 8-12 Hz). c) Inspiratory time 50% (1:1). d) amplitude 15 cmH2O(the range 15-25 cmH2O) NHFOV will only be provided with piston/ membrane oscillators able to provide an active expiratory phase (that is, Acutronic FABIAN-III, SLE 5000, Loweinstein Med LEONI+, Sensormedics 3100A).

SUMMARY:
This will be a prospective, multi-center, two-arms,parallel, randomized, controlled trial with a superiority design,conducted in China. The investigators conduct this multi-centre, randomized, controlled trial to test the hypothesis that NHFOV is more effective than nCPAP in the treatment of respiratory distress syndrome (RDS) in infants with a gestational age of less than 28 weeks when used as a primary noninvasive ventilation (NIV) mode.

DETAILED DESCRIPTION:
Preterm infants are eligible to the study if they they match the following inclusion criteria: (1) Gestational age between 240/7 and 286/7 weeks; (2) diagnosis of RDS. The diagnosis of RDS will be based on clinical manifestations (tachypnea, nasal flaring and or grunting) and a fraction of inspired oxygen (FiO2) greater than 0.25 for target saturation of peripheral oxygen (SpO2) 89% to 94%;; (3) Age less than 2 hours; (4)Informed parental consent has been obtained.

Neonates will be randomized and assigned either to nCPAP or NHFOV arms with a 1:1ratio, when patients fulfill all inclusion criteria. Randomization cannot be done earlier. Simple randomization will be done according to a computer-generated random number table and will be posted in a specific secured website 24/7 available. Twins will be allocated in the same treatment group. Infants randomized to one arm cannot crossover to the other or vice- versa during the study. For all the groups, if the fraction of inspired oxygen (FiO2) requirement is persistently higher than 0.30 per target SpO2 89-94% after starting the respiratory support, newborns receive Surfactant by "LISA" technique, administration of surfactant (Curosurf,Chiesi Pharmaceutics, Parma, Italy) 200 mg/kg.

After the administration of surfactant, if FiO2 requirement is persistently >0.4 to keep SpO2 89-94% or severe apnea episodes are present (defined as recurrent apnea with >3 episodes/h associated with heart rate <100/min or a single episode of apnea requiring bag and mask ventilation within a 24-hour period ) or at the blood gas (arterial or free-flowing capillary blood) PaCO2>60 mmHg and potential of hydrogen (pH)<7.20 obtained at least 1 hour after commencement of the assigned treatment, newborns are intubated and mechanically ventilated.

For all the newborns enrolled in the study, arterial or free-flowing capillary blood gas is checked every 6-12 hours, a cerebral and cardiac ultrasound screening is performed within 24 hrs. Further controls follow the routine of the ward.

ELIGIBILITY:
Inclusion Criteria:

(1) Gestational age between 240/7 and 286/7 weeks; (2) diagnosis of RDS. The diagnosis of RDS will be based on clinical manifestations (tachypnea, nasal flaring and or grunting) and a fraction of inspired oxygen (FiO2) greater than 0.25 for target saturation of peripheral oxygen (SpO2) 89% to 94%；（3） Age less than 2 hours

Exclusion Criteria:

* Intubated forany reasons at birth

  * Major congenital malformations or known complex congenital heart disease
  * No parental consent

Ages: 0 Hours to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, PhD, Study Chair — Children's Hospital of Chongqing Medical University
Locations (3):
- China (3):
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Qujing Maternity and cChild Healthcare Hospital, Qujing, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
URL: http://nasone.rxdemo.cn/admin/login/login

REFERENCES:
- [Derived] Li Y, Zhu X, Li LJ, Chen L, Yang Q, Xu L, Liang W, Lin X, Li C, Xue J, Liu L, Pan X, Ju R, Peng X, Tang W, Shi Y; NHFOV study group. Non-invasive high frequency oscillatory ventilation for primary respiratory support in extremely preterm infants: multicentre randomised controlled trial. BMJ. 2025 Oct 6;391:e085569. doi: 10.1136/bmj-2025-085569. PMID 41052898
- [Derived] Li Y, Zhu X, Shi Y; Noninvasive High-Frequency Oscillatory Ventilation Study Group. Non-invasive high-frequency oscillatory ventilation versus nasal continuous positive airway pressure in extremely preterm infants with respiratory distress syndrome: study protocol for a multicentre randomised controlled, superiority trial. BMJ Open. 2023 Mar 3;13(3):e068450. doi: 10.1136/bmjopen-2022-068450. PMID 36868587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August, 2022, through August, 2024, a total of 20 centers screened 729 infants, of which 405 were eligible. We recruited 360 infants (180 in each group), to account for dropouts. Finally, 342 infants completed the trial (170 in NHFOV; 172 in NCPAP group.)
Pre-assignment Details: 45 Did not undergo randomization 25 Refused to participate 11 transferr out of the NICU before randomisation 9 major congenital malformations
Period: Overall Study
Arm/Group | NCPAP | NHFOV
Started | 180 | 180
Completed | 172 | 170
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NCPAP | NHFOV | Total
Number analyzed (Participants) | 172 | 170 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 172 | 170 | 342
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: hours] | 1 (0.2) | 1 (0.3) | 1 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 74 | 142
  Male | 104 | 96 | 200
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 172 | 170 | 342
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 172 | 170 | 342
Birth weight [Mean (Standard Deviation); unit: g] | 970 (212) | 940 (204) | 950 (205)
Gestational age [Mean (Standard Deviation); unit: weeks] | 26.9 (1.2) | 27.0 (1.0) | 27.0 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure Within 72 Hours After Randomization 72 Hours After Randomization Need for Invasive Mechanical Ventilation
Description: The respiratory support failure will be considered if one of the following occurs: (1) severe respiratory acidosis (defined as PaCO2 >60mm Hg with pH<7.2) for at least 1hour; (2) hypoxia refractory to study intervention (defined as SpO2 <90%, with FiO2=0.4 and maximal pressures allowed in the study arm) for at least 1 hour after the administration of surfactant; (3) severe apnoea (defined as recurrent apnoea with >3 episodes/hour associated with heart rate <100/min or a single episode of apnoea requiring bag and mask ventilation) and (4) attending physician determined that urgent intubation is necessary.
Time Frame: within 72 hrs from the beginning of the study mode
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 48 | 27

2. Secondary Outcome: Rate of Airleaks(Pneumothorax and/or Pneumomediastinum) Occurred During Noninvasive Respiratory Support
Description: the diagnosis a Chest XR
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 4 | 1

3. Other Pre Specified Outcome: Rate of Bronchopulmonary Dysplasia
Description: defined according to the NICHD definition
Time Frame: 36 weeks of postmenstrual age
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 77 | 65

4. Other Pre Specified Outcome: Rate of Retinopathy of Prematurity (ROP)≥ 2nd Stage
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 39 | 40

5. Other Pre Specified Outcome: Rate of Necrotizing Enterocolitis (NEC) ≥ 2nd Stage
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 13 | 23

6. Other Pre Specified Outcome: Rate of Intraventricular Hemorrhage ≥ 3nd Grade
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 16 | 15

7. Other Pre Specified Outcome: Rate of Thick Secretions Causing an Airway Obstruction
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 10 | 12

8. Other Pre Specified Outcome: In-hospital Mortality
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 12 | 9

9. Other Pre Specified Outcome: Rate of Nasal Trauma
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 9 | 5

10. Other Pre Specified Outcome: Composite Mortality/BPD Tality/BPD
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 89 | 74

11. Other Pre Specified Outcome: Weekly Weight Gain
Description: in grams/d
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Mean (Standard Deviation); unit: g/Kg/day
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
g/Kg/day | 17 (6) | 16 (7)

12. Other Pre Specified Outcome: Overall Duration of Non Invasive Respiratory Assistance
Time Frame: the first 4weeks of life or until NICU discharge, whichever comes first
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
days | 27 [16 to 42] | 24 [14 to 43]

13. Other Pre Specified Outcome: Overall Duration of Hospitalisation
Time Frame: up to 2 years from birth
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
days | 57 [41 to 73] | 55 [41 to 75]

14. Other Pre Specified Outcome: the Rate of Patent Doctus Arterious
Description: If a pharmaceutical or surgical treatment is required is considered. Small doctuses closing spontaneously during the first days of life are not included.
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | NCPAP | NHFOV
Number analyzed (Participants) | 172 | 170
Participants | 32 | 35

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | NCPAP | NHFOV
All-Cause Mortality (participants affected / at risk) | 12/172 | 9/170
Serious Adverse Events (participants affected / at risk) | 0/172 | 0/170
Other Adverse Events (participants affected / at risk) | 0/172 | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05141435/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT05141435/ICF_001.pdf